CLINICAL TRIAL: NCT07251257
Title: The Seafarers' Continuous Glucose Monitoring Systems Study
Acronym: (SeaGM)
Status: Recruiting | Type: Observational
Sponsor: University of Surrey (Other)
Collaborators: The UK Maritime and Coastguard Agency (Unknown)
Responsible Party: Sponsor
Other Study IDs: FHMS 23-24 062 EGA/ERM ID 2469; #1716 (Other Grant/Funding Number: Seafarers' Charity and Fishmongers Company in UK)
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Insulin Dependent Diabetes
Keywords: insulin dependent diabetes; Continuous glucose monitoring; Seafarers; Fishers
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Seafarers wearing CGM device: Fifty seafarers will be recruited to participate in a one-year study utilizing the Dexcom G7 Continuous Glucose Monitoring (CGM) system.
  Participants will also be enrolled in the web-based Fishers Watch application, which will deliver daily reminders via text message prompting them to note on their activities both at sea and on land.

SUMMARY:
People with diabetes sometimes consider that they are subjected to unfair discrimination in the occupational or work environment. These include safety-critical activities, such as operating machinery and driving 1-3. Some occupations preclude the use of medications that lower blood glucose, particularly insulin. Safety regulators, occupational health physicians and national organisations frequently have to balance the competing priorities of individual rights against public safety.

Modern treatment, with advances in insulin therapy and glucose monitoring, combined with rigorous clinical assessment and review, has allowed stereotypical attitudes to be challenged and advocated individual assessment with respect to safety criteria. Along with the UK Driving and Vehicle Licensing Agency (DVLA) and Civil Aviation Authority (CAA), the Maritime and Coastguard Agency (MCA) have accepted that insulin-treated diabetes should not be an absolute contra-indication to partaking in these occupational activities4. However, as the Disability Discrimination Act (1995) recognises that there may be specific employment-related hazards, fitness to work should be assessed on an individual basis. Therefore, each of these transport agencies has established regulatory standards for their respective domains, with the priority of minimising hypoglycaemic incapacitation risks. The CAA, for example, has worked alongside other European countries to use the ARA.MED.330 protocol and require medically certified pilots to check their blood glucose levels regularly before and during flights. In 2010, the UK CAA's expert committee reviewed the knowledge and policies concerning flying and it was decided that Continuous Glucose Monitoring (CGM) systems were not accurate enough and instead used finger prick-blood glucose monitoring (SMBG) as the gold standard. Since then, the protocol has been successfully implemented and there are current works in progress that demonstrate sufficient accuracy in modern CGMs as a viable alternative to SMBG.

Similarly, the guidelines devised by the MCA, Approved Doctor's Manual (ADM), place a great emphasis on the type and treatment of diabetes, with the primary concern being risks of cognitive impairment or incapacitation5. Emphasis is placed on the need for able glycaemic control and "full awareness of impending hypos, with no reported or observed significant hypoglycaemic episodes in the last year". The guidance stipulates that certification may be restricted on individuals pending their medication side effects, compliance, and vascular risk factor control. Previous regulations prevented seafaring individuals such as insulin-treated seafarers from partaking in lone watchkeeping/lone-working roles and restricted them to near-coastal duties (150-200 nautical miles) (Appendix 1). Current regulations allows for exemptions for certain vessels, provided that the seafarer's diabetes control remains stable and is subject to blood glucose monitoring. Regardless, an approved medical assessor is needed to conduct these specific medical assessments in line with the statutory standards in MSN 1886 and guidance in the ADM.

All seafarers who are insulin-dependent and licenced to undertake seafaring in the UK will be invited to participate in this study.

DETAILED DESCRIPTION:
STUDY DESIGN and METHODS of DATA COLLECTION AND DATA ANALYSIS This will be an observational and feasibility study on the use of the insulin-treated fisher seafarers' with or without own real-time CGM systems, such as Dexcom G6®, Dexcom G7®, Guardian 4 or Abbott Freestyle Libre. The participating seafaers with insulin-treated diabetes who are currently monitoring their glucose levels using a CGM and certified to undertake commercial work at sea and will be taking corrective actions according to their glucose readings. The CE marked Dexcom G7® will be provided to the participants in the study for 1 year. A questionnaire is designed to streamline the process of the glucose management while at sea. Additionally, a progressive web app (Fishers Watch) will be provided and accessible by participants via their own smartphone devices to enable better recording of adverse/diabetes-related events and activities during the study and can also help indicate their on- and off-duty periods to facilitate data analysis.

Participants will be encouraged to use their CGM glucose measurement data from their own devices, to assist with their diabetes management. The involvement of the participants in the study will be 12 months. The participants will be reminded during the study that it is crucial to log their CGM glucose measurements alongside their activities and any hypoglycaemic/hyperglycaemic episodes within this timeframe.

Screening/run-in period Seafarers will be recruited via the MCA ML5 or ENG1 medical certification processes for medical certification (see Appendix 2). All insulin treated seafarers who presenting for an ML5 or ENG1 certificate who are assessed as fit to work at sea will be asked for and will be provided with information and a consent form for the Scheme6 (Appendix 3). All signed consent forms confirming to be approached by the investigators at the University of Surrey, will be forwarded to the investigators at the University of Surrey. We, the investigators at Surrey, will then have the email contact for the seafarer and we can then approach the interested seafarers directly (Appendix 1 Supplementary Material 2).

Screening visit (Virtual visit 1)

All seafarer will be invited for a virtual/online/phone screening visit. The virtual meetings will be held on TEAMs.

Before screening takes place, participants (seafarers) will be provided with verbal and written information about the trial and the procedures involved in a virtual visit with prior appointment. They will be fully informed of their responsibilities and rights while participating in this exploratory trial. They will be given the opportunity to ask questions and ample time to consider participation. Participants who wish to participate in the trial will be required to sign and date an Informed Consent Form prior to any trial-related activities taking place. All participants will be provided with a copy of fully signed and dated Informed Consent Form.

The following information will be recorded from the annual diabetes clinic visit at the GP: health data: medical history, concomitant medication, and HbA1c results and DOB, age, tobacco smoking status, alcohol intake. The subject will be asked to share the data with the PIs in the study for the clinical report files (CRF) files. If the participant fulfils all inclusion criteria and none of the exclusion criteria they will be accepted into the study.

Visit 1 On TEAMs:

Following screening, seafarers who are eligible for the study will be recruited in this virtual visit on TEAMs by the University of Surrey investigators. The participants will be informed that they will be required to monitor their glucose levels using their own the study CGM device at all times during the next 12 months of the study and make their electronic glucose records available to the research team through the Dexcom Clarity platform. The participants will be asked to record any out-of-range glucose measurements and any events or consequences when they are at sea. This data will be collected using a dedicated progressive web-app designed for this study (Fishers Watch web-app). The participants will also record the dates they at sea at sea and when working at sea or at rest.

A questionnaire will be distributed to all eligible participants to ensure the proposed usage of devices will be compatible with their work activities while at sea. This questionnaire will be used to evaluate the impact of this study on their work and to inform on further changes to the protocol as necessary.

The participants will be supplied with Dexcom G7® CGM sensors sufficient for the next 6months. The supplies will be sent by post.

Virtual Visit 2 on TEAMs: This will take place months after virtual visit 1 (3 months±7 days).

Participants are reviewed virtually/online on TEAMs at 3 months. They will be asked if they are willing to continue with the study participation. If they decide not to take part, we will let the Medical team at the MCA agency know of their decision. The adverse events and concomitant medications will be reviewed and recorded: The data from their study CGM will be reviewed and collected from Dexcom Clarity platform. The events and activities recorded by the participants' in the Fishers Watch App between visit 1 and visit 2 will also be collected.

As in virtual visit 1, the participants will be asked to record any out-of-range glucose measurements and any events or consequences when they are at sea. This data will be collected using the Fishers Watch App for the period between virtual visit 2-visit 3.

Virtual Visit 3 on TEAMs: This will take place 6 months after visit 1 (6 months±7 days).

Participants are reviewed virtually/online on TEAMs at 6 months. They will be asked if they are willing to continue with the study participation. If they decide not to take part we will let the Medical team at the MCA agency know of their decision. The following will be reviewed and recorded: adverse event, concomitant medication. The data from their study CGM will be reviewed and collected from Dexcom Clarity platform. The events and activities recorded in the participants' Fishers Watch App between visit 2 and visit 3 will also be collected.

As in visit 2, the participants will be asked to collect the data from their CGM in the study Fishers Watch App for the period between virtual visit 3-visit 4.

The participants will be supplied with Dexcom G7® CGM sensors sufficient for the next 6months. The supplies will be sent by post.

Visit 4 (End study): This will take place 12 months after visit 1 (12 months ± 7 days).

Participants will be asked to attend the virtual appointment 6 months after visit 3. They will be asked if they are willing to continue with the study participation. The following will be reviewed and recorded: adverse event, concomitant medication, HbA1c required for the annual diabetes clinic at the GP. The data from their CGMS will be collected and reviewed from Dexcom Clarity platform. The events and activities recorded in the participants' the Fishers Watch App between virtual visit 3 and visit 4 will also be collected.

Measurements (recordings):

Virtual Visits 1 and Visit 4 Participant's HbA1c measurements will be retrieved from their most recent medical records at Visit 1 and Visit 4.

CGM Data collection:

Virtual Visits 1, Visit2, Visit 3 and Visit 4

Data from the participants' CGM system (via Dexcom Clarity) and the Fishers Watch App for the periods between virtual visit 1- visit 2, visit 2-visit 3 and visit 3-visit 4 will be collected.

DURATION OF STUDY PARTICIPATION

* Duration of study participation for each patient - 12 months

PATIENT SAFETY SAFETY ENDPOINTS ASSESSED IN THIS STUDY

* Clinical safety
* Adverse event collection

SAFETY INSTRUCTIONS

* Self-measured capillary blood glucose
* Hypoglycaemia
* Local tolerability
* Allergic or allergic-like reaction

ADVERSE EVENT REPORTING Any adverse events will be reported to the Sponsor within 72 hours of becoming known to the research team. The MCA has agreed to inform the research team when made aware of any seafarers' adverse health events, including any injuries as a result of deranged glucose levels

ANNUAL SAFETY REPORTING and END of STUDY REPORTING

At the end of the year from the initiation date of the study, an annual report will be submitted to the University Ethics committee. At the end of the study, an end study report with all the data will also be submitted to both the Sponsor and the University Ethics Committee.

Participants will be withdrawn from the study by investigators if:

1. Participants experience an adverse reaction to the sensor (e.g. severe allergic reaction or intolerance)
2. The participant develops a medical condition either prior to entering or during the study, which may compromise their safety during free-living or seafaring activities and/or adversely and affect the outcome of the study.
3. The participant is consistently non-compliant.

   Unless the participant specifically requests that their data is not used, all data prior to subject withdrawal will be used in analysis, however the deadline for withdrawal will be 7 days following completion of the study, as this is when statistical analysis will be completed.

   Data analysis methods
   * Data collected from visit 1, visit 2, visit 3 and visit 4 and further data from the participants' logbooks will be transcribed by the PI responsible at the MCA site.
   * The CGMS/Flash data will be held on the readers and on the cloud, a copy of which will be sent to the PI and the investigators at the University of Surrey.
   * Data per participant will be coded and anonymized using SeaGM 001 to SeaGM 050.
   * Glucose variability on land before departure and during their time at sea
   * The variability in normal living and the time in and out of range will be calculated using the data from the CGM/Flash devices, collected by the PI.
   * The data from Fishers Watch web-app will be downloaded and saved by the PI and the investigators at the University of Surrey on the University computer as excel files for participants SeaGM 01 to SeaGM 50.
   * Questionnaire data will be analysed.
   * Simple statistical analysis will be performed using SPSS and Excel.

   ANALYSIS POPULATIONS

   • Efficacy populations - all patients who complete the 12 months study. There will be an interim analysis of the data at the 3, 6 and 12 months' time points.

   • Data will be stored only on the UK MCA or University of Surrey computers.

   • Data from the study will be archived at the University of Surrey.

   5 STUDY SETTING The seafarers in the UK are known to the UK Maritime & Coastguard Agency The address (105 Commercial Rd, Southampton SO15 1EG, United Kingdom), will be invited to take part in this study.

   • Protocol will be submitted for full ethical approval from the University of Surrey.

   • Participants will be accessed and invited to the study by the PI at the MCA site.

   • Insulin-treated seafarers attending a virtual medical assessment clinic as part of their certification requirement once a year, so the setting of this study fits with their usual clinic visits, with two extra virtual visit at 3 &6 months to ascertain the feasibility of the protocol.

   • Once the seafarers consented to be contacted by the investigators at the University. The investigators at the university will then organise the Virtual/phone screening visit 1 and the following 3 virtual visits 2, 3 and 4.

   • The TMF and copies of consent forms will be kept at the Leggett building at the University of Surrey

   6 SAMPLE AND RECRUITMENT 6.1 Eligibility Criteria NUMBER OF PATIENTS PLANNED: Fifty seafarers with insulin-treated diabetes who are also certified for commercial maritime activities.

   6.2 Sampling

   6.2.1 Size of sample This is the first study of glucose variability in this population of seafarers; however, sample size was based on the primary endpoint of continuous glucose monitoring during 24 hour period. This is a unique population and this observational study will provide informative data. The previous studies of participants with type 1 diabetes, adequate data was produced to calculate variability and data out or range for glucose concentration during work/flight periods7. The participants acted as their own controls, increasing the power for analysis. The correlation between measurements in the same person is unknown so this was assumed to be zero (the worst-case scenario). Completing the study in 50 seafarers patients would have the power of 80% to detect a difference of 20% which would be considered clinically significant.

   6.2.2 Sampling technique The study population is self-selecting (those with insulin-treated diabetes and certified to undertake commercial maritime activities).

   6.3 Recruitment The study population is self-selecting (those with insulin-treated diabetes and certified to undertake commercial maritime activities). The PIS will be sent to the participants at least 24hours prior to the virtual screening visit with the University of Surrey Investigators.

   6.3.1 Sample identification The PI at the MCA site will identify the participants from the MCA clinic records.

   There will be no payments to the participants.

   6.3.2 Consent

   A letter/email of invitation will be sent to the eligible seafarers. Informed consent will be obtained prior to the participant undergoing any activities that are specifically for the purposes of the study.

   6.3.2 Withdrawal of Consent The participants can withdraw their consent at any time. The data collected up to withdrawal will be used in the analysis.

   7 ETHICAL AND REGULATORY CONSIDERATIONS The simple observational study does not involve any NHS organisation and will therefore be submitted to the University of Surrey research ethics committee.

   7.1 Assessment and management of risk The CGM and Flash devices are allowed in the patient population and therefore there are no additional risks in the study.

   The visits are held virtual.

   7.2 Research Ethics Committee (REC) and other Regulatory review Before the start of the study, a favourable opinion will be sought from the University Ethics Committee (UEC)

   Regulatory Review & Compliance The PIC site and where the study will take place are not NHS sites, however, the study will comply with GCP. The PI at the site will provide a CV and GCP training certificate to the University Ethics Committee (UEC).

   7.3 Peer review This is an investigator-led study and has been through rigorous peer review at MCA and has been deemed high priority study likely to lead improved scientific understanding.

   7.4 Patient & Public Involvement

   • N/A

   7.5 Protocol compliance Protocol compliance will be obvious due to the nature of the study and collection of the data from the CGM/Flash monitoring systems. Virtual Visit 2 is designed to find out the compliance and workability of the designed protocol. (If there are gaps in the data collection this will be easily picked up on the monitor. No data or gaps in the data collection will mean one scenario of the following: non-compliance, sensor not on properly, no connection between the sensor and monitor over a long period over 6 h or no charge in the monitor).

   The logbook data or the data entered by the seafarers into the Fishers Watch App is also important if this was filled in poorly that would be considered non-compliance. The non-compliance will be reported to the PI at the MCA.

   7.6 Data protection and patient confidentiality All Data will be anonymised before data analysis and will be compliant with the requirements of the Data Protection Act 2018 (GDPR).

   The study PI and the research team will ensure that the participants' anonymity is maintained. Once a consent form has been signed the participant will be given a study identification number. The participants will be identified only by participants ID number in their clinical research forms (CRF) and any electronic database. The hard copies of the anonymised Research data will be kept in a locked cupboard, in room 21PG00 at the Leggett Building University of Surrey. All documents will be stored securely and only accessible by study staff and authorised personnel. The study will comply with the Data Protection Act, which requires data to be anonymised as soon as it is practical to do so. The hourly glucose concentration data entered by the participant is uploaded to the external system, called the Fishers Watch and will be deleted as soon as the data is transferred to the UoS systems. The system will have the participant's smart mobile number however no other data will be accessed by the system. The Data Protection Officer at the University of Surrey has been approached and the vendor assessment completed. The assessment deems the vendor (Patient Watch Ltd., Company Number 14114586) of low risk.

   The data from the CGM/Flash systems will be collected continuously. The at-sea incidents and comments entered by the participant are uploaded to the external system of Fishers Watch progressive web app. Glucose measurements are routinely uploaded to CGM device manufacturers' systems throughout the world. Data will be collected in compliance with GDPR (2018) and the system has been approved by the Royal Surrey Data Protection Impact Assessment.

   Access to identifiable data that is name, address, date of birth, telephone number, next of kin, GP name and address, will be limited to selected members of the research team and to regulatory authorities, the Sponsor, and the host organisation for auditing and monitoring purposes. This information and other personal details will not be included in analysis, or in publications or reports. All information collected during the study will be identified by a unique code so that the participant cannot be identified. All data will be kept on secure MCA or University of Surrey computer servers and in a secure office environment within the MCA and University of Surrey.

   The researchers will use the password protected folder in the shared drive at the University of Surrey in the following folder address: S:\Shared_Projects\PG00_PGMS_Mass_Spec_Lab to save the documents and data from the study which will be accessible to all in the research team.

   All project data related to the administration of the project, (e.g. consent form) will be held for at least 6 years and all research data for at least 10 years in accordance with University policy. The personal data will be held and processed in the strictest confidence and in accordance with current data protection regulations.

   The PI will be the data custodian.

   7.7 Indemnity and Insurance The study falls within the terms and conditions of the University research policy. The Sponsor will not take out a specific insurance cover for this study.

   7.8 Access to the final study dataset All investigators will have access to the pseudonymised data set.

   8 DISSEMINIATION POLICY 8.1 Dissemination policy

   It is likely this study will be presented at scientific international peer reviewed meetings and ultimately published in a peer reviewed scientific journal but only in the form of average values for the group; no individual subject data will be published or presented in scientific meetings.

   8.2 Authorship eligibility guidelines and any intended use of professional writers The authors will be those with substantial input to the design and implementation of the study. This will include the PIs and co investigators. No professional writers will be involved in the design or publication of this study.

ELIGIBILITY:
Inclusion Criteria:•

* Any ethnicity
* Seafarers requiring insulin replacement therapy,
* Holding a valid ML5 or ENG1 certificate
* Able and willing to wear a Continuous Glucose Monitoring system (GCMS) for 12 months
* Able and willing to document out of range glucose values and activities in Fishers Watch App a while at sea

Exclusion Criteria:

* Outside of the stated age range.
* Not able to use using a CGM glucose monitoring system for monitoring the glucose levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seafarers requiring insulin replacement therapy, and holding a valid ML5 or ENG1 certificate
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the glucose monitoring of CGM systems in the context of their usual occupational activities and establish its feasibility as a routine glucose monitoring device while at sea. | 12 months
  Evaluation of the glucose monitoring of CGM systems in the context of the seafarers' usual occupational activities and establish its feasibility as a routine glucose monitoring device while at sea. Glucose measurements will be based on a traffic light system, with <5 mmol/L coded as red, 5-20 mmol/L as green, and >20 mmol/L coded as red as per our maritime protocol.

SECONDARY OUTCOMES:
Glucose variability while working or on rest period at sea | 12 months
  Glucose variability while working or on rest period at sea
Time in and out of range while seafaring (targets used as other clinical trials) | 12 months
  Time in and out of range while seafaring (targets used as other clinical trials)
Feasibility and safety assessment of using CGM systems during seafaring activities | 12 months
  Glucose variability while at sea in comparison to on land
Questionnaire data an overview of participants' preferences | 12 months
  Questionnaire data will provide an overview of participants' preferences towards glucose monitoring devices and their trust in the systems used to manage their glucose levels.

CONTACTS AND LOCATIONS:
Overall Officials: David L Russell-Jones, MD, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey FHMS Nutritional Sciences, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garden GL, Hine JL, Mitchell SJ, Hutchison EJ, Gaffney TP, Hofmann V, Frier BM, Shaw KM, Heller SR, Koehler G, Roberts GA, Russell-Jones DL. An Evaluation of the Safety of Pilots With Insulin-Treated Diabetes in Europe Flying Commercial and Noncommercial Aircraft. Diabetes Care. 2020 Dec;43(12):2923-2929. doi: 10.2337/dc20-0277. Epub 2020 Jun 25. PMID 32586987
- [Result] Ehrmann D, Heinemann L, Freckmann G, Waldenmaier D, Faber-Heinemann G, Hermanns N. The Effects and Effect Sizes of Real-Time Continuous Glucose Monitoring on Patient-Reported Outcomes: A Secondary Analysis of the HypoDE Study. Diabetes Technol Ther. 2019 Feb;21(2):86-93. doi: 10.1089/dia.2018.0332. Epub 2019 Jan 7. PMID 30615479
- [Result] Wadwa RP, Laffel LM, Shah VN, Garg SK. Accuracy of a Factory-Calibrated, Real-Time Continuous Glucose Monitoring System During 10 Days of Use in Youth and Adults with Diabetes. Diabetes Technol Ther. 2018 Jun;20(6):395-402. doi: 10.1089/dia.2018.0150. Epub 2018 Jun 14. PMID 29901421
- [Result] Shah VN, Laffel LM, Wadwa RP, Garg SK. Performance of a Factory-Calibrated Real-Time Continuous Glucose Monitoring System Utilizing an Automated Sensor Applicator. Diabetes Technol Ther. 2018 Jun;20(6):428-433. doi: 10.1089/dia.2018.0143. PMID 29923775
- See also: Maritime & Coastguard Agency. Approved Doctor's Manual Seafarer Medical Examinations. 2020;1886. — https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/901465/Approved_Doctors_Manual_July_2020.pdf
- See also: Maritime & Coastguard Agency. MSN 1883 (F) Amendment 5 Work in Fishing Convention (No. 188): Medical examination and certification for fishers [Internet]. 2024. — https://www.gov.uk/government/publications/msn-1883-f-amendment-5-work-in-fishing-convention-no-188-medical-examination-and-certification-for-fishers/msn-1883-f-amendment-5-work-in-fishing-convention-no-188-medical-examination-and-certification-for-fishers